CLINICAL TRIAL: NCT06819995
Title: Accuracy of Static Guided Implant Surgery: 3D-printed vs Milled Surgical Guides, a Randomized Clinical Trial
Brief Title: Accuracy of Static Guided Implant Surgery: 3D-printed vs Milled Surgical Guides
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Complutense de Madrid (Other)
Collaborators: Klockner Implant System (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 24/716-EC_X
Record Dates: First submitted 2024-12-04; First posted 2025-02-11 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2024-12

CONDITIONS: Dental Implant; Guided Surgery Accuracy
Keywords: Dental implant; Guided surgery; Surgical guide; 3D printing; Milling

STUDY DESIGN:
Intervention Model Description: Two-arm, double-blind (examiner, and patient), single-center parallel randomized controlled trial
Who Masked: Participant, Outcomes Assessor
Masking Description: Each patient will be randomized into the milled or 3D-printed group according to a balanced distribution system via a computer-generated table of random numbers. Allocation concealment will be kept during the surgery by means of opaque envelopes so that the patient is blinded, and it will be kept until the moment of data analysis by an independent researcher not involved in the execution of the clinical interventions. Opaque sealed envelopes will be opened at the milling center once the 3D implant planning has finished, been checked, and sent.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 3-D printed guide (Active Comparator): Patients will receive guided dental implants by means of a 3D-printed static surgical guide.
  Interventions: Procedure: Static guided implant placement with a 3D printed guide
- Milled guide (Experimental): Patients will receive guided dental implants by means of a milled static surgical guide.
  Interventions: Procedure: Static guided implant placement with a milled guide

INTERVENTIONS:
Procedure: Static guided implant placement with a 3D printed guide — 3D-printed guides (E-Guide resin, EnvisionTEC®, Germany) (D4K Pro printer, EnvisionTEC®, Germany) performed by acommercial manufacturing center (Archimedes, Spain). All guides will be designed with guide sleeves. Finally, the guide will be post-processed and sterilized according to the manufacturer's recommendations.
  Other Names: 3D-printed sCAIS
  Arms: 3-D printed guide
Procedure: Static guided implant placement with a milled guide — Milled guides (anaxCAM PMMA Clear blanks, Anaxdent, Germany) (CORiTEC 150i PRO miller, Imes-icore®, Germany). All guides will be designed with guide sleeves. Finally, the guide will be post-processed and sterilized according to the manufacturer's recommendations.
  Other Names: Milled sCAIS
  Arms: Milled guide

SUMMARY:
Dear Patient,

You are invited to participate in a clinical study. To understand the study, please carefully review the following information. If you have any questions, feel free to ask the dentist leading the study.

Dental implants are an effective, long-term solution for replacing missing teeth. They replace the root of a lost or unsalvageable tooth, supporting a crown or prosthesis to restore function and aesthetics. Proper placement is crucial for implants to function and last. Guided implant surgery is a technique that improves precision using customized surgical guides created from patient records, such as radiographs and scans. These guides act as templates to ensure accurate implant placement, optimizing functionality, aesthetics, and minimizing complications.

There are two main methods for fabricating surgical guides: milling, which cuts material into shape, and 3D printing, which builds material layer by layer. This study aims to evaluate the differences in accuracy and long-term outcomes between implants placed using guides created by these two methods. Both clinical results (appearance and function) and radiographic results (bone integration) will be assessed to determine the best method for guide fabrication.

You were selected for this study because you require dental implant rehabilitation. After clinical and radiographic evaluations, we determined you are a suitable candidate for implant placement to restore your dental function and aesthetics.

If you choose to participate, the following steps will be taken:

1. A thorough examination of your dental health, including radiographs and photographs.
2. Planning and guided surgery performed at the Postgraduate Program in Periodontics.
3. Random assignment to receive either a 3D-printed or milled surgical guide. This assignment will be computer-generated and remain unknown until the study concludes.
4. Surgery under local anesthesia, lasting 1-2 hours, followed by suture removal after 7 days and follow-ups at 2 and 3 weeks to monitor healing.
5. At 3 months, clinical and radiographic evaluations will be performed, and digital impressions will be taken to assess differences between planned and final implant positions. The impressions will also be used to fabricate your final prosthesis, which will be placed approximately one month later.
6. Follow-ups at 6 and 12 months after prosthesis placement will assess implant stability and overall outcomes. The study will conclude after this final evaluation.

Participation involves certain risks:

* Anesthesia-related risks, such as allergic reactions, prolonged numbness, or local tissue damage.
* Surgical risks, including pain, swelling, bleeding, infection, temporary or permanent numbness, and damage to adjacent teeth or roots.
* Implant failure, either during initial bone integration or later, requiring additional treatment or replanning.
* Risks of material failure, such as fractures or loosening of prosthetic components.

By participating, you will avoid costs for the implants, healing abutments, and surgical guides (approximate savings: €800-€1,200). However, you will be responsible for surgery (€60), prosthetic components (€250 each), and final restorations (€350 per crown). Participation also includes close monitoring of your implants for one year, allowing for early detection and management of complications at no cost.

Participation is voluntary. If you decide not to participate, it will not affect your care. You may also withdraw from the study at any time without penalty, although clinical follow-ups are recommended to monitor your treatment outcomes.

Your data will be handled anonymously and securely, in compliance with data protection laws (e.g., Spain's Organic Law 3/2018). Data will be used solely for research purposes and not for commercial gain. Identifiable information will not be published, and your rights to access, correct, or delete your data will be upheld.

If you have questions, you may contact the research team by phone or email. You may also consult your dentist or the Ethics Committee. A copy of this document is available for your records.

Thank you for considering participation in this study.

DETAILED DESCRIPTION:
1. SCIENTIFIC BACKGROUND AND RATIONALE

   Traditionally, implant placement has been based on bone availability, with the implant industry focused primarily on enhancing implant survival by increasing the chances of osseointegration. In contrast, the position of the final prosthetic rehabilitation was considered of secondary importance. In certain instances, this approach may result in biological, prosthetic, and aesthetic complications. In contemporary dentistry, evaluating the success of implant therapy transcends the mere evaluation of implant survival and involves a comprehensive assessment that takes into consideration the long-term stability of soft and hard peri-implant tissues, access for oral hygiene, aesthetic demands, occlusal and functional dynamics, implant loading potential, and minimal invasiveness.

   Digital-based planning and guided surgery can maximize the chances of placing implants in an ideal prosthetic position. Different types of guided surgery have been described in the literature: (1) Static cast-based partial guidance, which considers the final prosthetic position without considering bone morphology and in which bone bed preparation and implant placement are free-handed. (2) Static computer-based partial guidance, in which the underlying bone morphology is considered in manufacturing the surgical guide, and that can be used for the initial, partial, or complete osteotomy, but implant placement is still free-handed. (3) Static computer-based full guidance that entails the utilization of a pre-made surgical template, involving both complete osteotomy preparation and implant placement guided by a prosthetically driven surgical guide; and (4) Dynamic guidance, that allows real-time guidance during drilling, with the implant position dynamically displayed on computed tomography data. Dynamic guides are associated with higher economic costs and pose challenges in in their clinical implementation, and consequently, static guides are more frequently utilized. The type of support for the guide can be categorized into three groups: mucosal-supported, tooth-supported (may be combined with mucosal-supported), or bone-supported.

   Implant surgical guides can be produced through two manufacturing processes: subtractive and additive manufacturing. The subtractive approach involves milling the surgical guide from a larger polymer block through a computer-numeric controlled machine. The additive approach is based on 3D printing the guide by sequential layering. In general, additive processes are more frequently employed, due to reduced expenses, the production of more guides per printing session, and minimal waste.

   Recent systematic reviews have demonstrated that static fully guided surgery has higher accuracy to achieve the planned position than free-handed and partially guided implant placement . Indeed, different RCTs have reported higher chances of obtaining a prosthetically correct implant position allowing for screw-retained restorations, lower mean depth deviation, lower angular deviation, as well as three-dimensional body deviations when using static guidance with respect to free-handed implants.

   However, there is no conclusive evidence on the differences in accuracy when comparing static guides fabricated either through an additive or a subtractive process.
2. STUDY OBJECTIVES The primary aim of this study is to determine whether there are any differences on the accuracy of implant placement using two different types of static surgical guides: 3D-printed vs. milled. The null hypothesis is that there will be no differences in the accuracy of implant placement when comparing 3D-printed and milled surgical guides.

   The primary objective of this investigation will be to evaluate the accuracy of implant placement defined in terms of differences in precision and trueness (ISO 5725-2) between the planned and the final implant position, when comparing 3D-printed and milled surgical guides.

   As secondary objectives the following outcomes will be evaluated: peri-implant health outcomes (bleeding on probing, suppuration, probing depth), plaque index, implant survival, implant success, surgery-related outcomes (time, difficulty [VAS scale], and wound healing index), and patient-reported outcomes measures.

   2.1 Clinical relevance A correct implant position is important for the long-term success of implant therapy. Static computer-assisted implant placement is an alternative to free-hand surgery that has shown higher accuracy in reaching an appropriate implant position. However, data on the accuracy associated to the use of either milled or 3D-printed implant surgical guides is limited.
3. MATERIALS AND METHODS

3.1. Study design Two-arm, double-blind (examiner, and patient), single-center parallel randomized controlled trial.

3.2. Trial centers This study will be carried out in the clinic of the Postgraduate of Specialization in Periodontology and Implant Dentistry at the Complutense University of Madrid (Spain)

3.4. Intervention / Study Procedures 3.4.1. Screening and Baseline Procedures All potential study participants will be screened for eligibility according to the inclusion and exclusion criteria and will be informed about the study procedures.

3.4.2. Informed Consent Written informed consent must be obtained from each patient prior to performing any study procedure or assessment. Before enrolling a subject, the Investigator will explain the study protocol, procedures, and objectives to the subject and/or legal guardian or legally authorized representative. When the subject understands and is willing to participate in the clinical trial, he/she must sign and date the IRB-approved Informed Consent Form (ICF). The ICF describes the study and the potential discomforts, risks, and benefits of participating. One copy of the consent form will be provided to the subject, and one copy will be maintained with the subject's permanent medical records. The study site personnel must also enter the date the informed consent was signed in the subject's source documentation or medical record.

3.4.3. Randomization Each patient will be randomized into the milled or 3D-printed group according to a balanced distribution system via a computer-generated table of random numbers. Allocation concealment will be kept during the surgery by means of opaque envelopes so that the patient is blinded, and it will be kept until the moment of data analysis by an independent researcher not involved in the execution of the clinical interventions. Opaque sealed envelopes will be opened at the milling center once the 3D implant planning has finished, been checked, and sent.

3.4.4. Pre-study phase and guide fabrication Upon inclusion in the study, all potentially eligible patients (all patients meeting primary inclusion criteria) will receive oral hygiene instructions (OHI) according to their individual needs. Patients with residual dentition with signs of periodontitis will also receive periodontal therapy.

After this, all eligible patients will be re-evaluated according to their compliance with oral hygiene procedures (secondary exclusion criteria) to establish their inclusion in the trial.

* A preoperative intraoral scan of the receptor arch and a cone-beam computed tomographic scan of the arch of interest will be acquired to digitally plan implant placement. A blinded investigator with experience in implant dentistry will perform the virtual planning for all cases based on a prosthetic-driven implant position using the Medconnect software platform (Archimedes).
* The digital planning will consist of 3-dimensional radiographical measurements on DICOM data to assess the optimal position of the implant(s) based on digital wax-up. An STL file will be used to construct the surgical guide (S0). At this stage, if additional bone regeneration procedures are needed to achieve the ideal position of the implant(s), the surgical planning will be aborted, and other options will be offered to the patient. Transalveolar sinus floor elevation up to 2 mm will be allowed. The surgical guide will be designed aiming primarily for tooth support or mixed (tooth and mucosal) support. Cases where this cannot be achieved will be excluded.
* Once this process has ended, patients will be randomized as described previously to receive milled guides (anaxCAM PMMA Clear blanks, Anaxdent, Germany) (CORiTEC 150i PRO miller, Imes-icore®, Germany) or 3D-printed guides (E-Guide resin, EnvisionTEC®, Germany) (D4K Pro printer, EnvisionTEC®, Germany) performed by the same commercial manufacturing center (Archimedes, Spain). All guides will be designed with guide sleeves.
* Finally, the guide will be post-processed and sterilized according to the manufacturer's recommendations.
* Before the day of surgery, the surgical guides will be tested for fit and stability through tactile inspection. In poorly fitted guides, new intraoral and CBCT scans will be obtained to repeat the digital planning phase.

3.4.5. Surgical procedure

* All implant surgeries will be performed under local anesthesia by one of five calibrated, experienced surgeons who have not been involved in the digital planning of the implant position.
* All implants will be bone-level Klockner Vega® implants (Klockner Implant System, Spain), ranging from 3.5 to 4.5 mm in diameter and 8 to 12 mm in length.
* The selection of performing a flapless or a full thickness mucoperiosteal flap will be determined before surgery by measuring the availability of keratinized mucosa. A flapless technique will be selected for cases where at least 2mm of surrounding keratinized mucosa can be ensured around the whole implant. If performing a flap, a crestal design will be used to assure that at least 2 mm of keratinized mucosa is left on the buccal and lingual flaps.
* Implant bed preparations and insertions will be done through the 3D surgical guides following the manufacturer's protocol (Sniper Guide System, Klockner Implant System, Spain). All implants will be placed 1-1.5 mm subcrestally.
* A transmucosal healing abutment and interrupted non-resorbable 5/0 sutures will be placed.

3.4.6. Postoperative care Patients will be instructed to rinse postoperatively for 1 min with 0.12% CHX + 0.05% CPC (Perio-aid treatment®) three times a day for 2 weeks. Patients will also be allowed to take Ibuprofen 600mg every 8 hours as needed. If necessary, Paracetamol 650mg will be intercalated. Patients will be asked to keep a record of the medication taken (type of medicine, frequency, and number of days).

Patients will be instructed to refrain from performing regular oral hygiene in the surgical area immediately after the surgery for one week. Smokers will be asked to limit (and possibly quit) smoking to no more that 5 cigarettes per day.

Sutures will be removed after 7 days, and self-performed biofilm control in the surgical area will be reinstituted with the use of a soft toothbrush. At one month, patients will be instructed to start routine self-performed oral hygiene procedures and will receive supragingival polishing with an air polishing device (Airflow® EMS) and a subgingival non-abrasive powder (Erythritol, Plus Powder®, EMS).

Three months after surgery, digital impressions will be taken at the implant level for single unit restorations or at the abutment level (Permanent) for multiple unit restorations. If intermediate abutments are used, the day of digital impression will be screwed and not removed anymore. Titanium bases will be used to cement zirconia CAD-CAM restorations at the laboratory, which will be then screw at the implant or the abutment the day of loading. To standardize the prosthetic designs, all the restoration will be fabricated at the same laboratory (Symmetrya, Oporto). Functional loading will be considered as the baseline visit for the subsequent follow-up. Professional prophylaxis and OHI will be performed at 6 and 12 months using ultrasonic and air polishing devices (Prophylaxis Airflow Master Piezon® EMS) and a subgingival non-abrasive powder (Erythritol, Plus Powder®, EMS).

3.4.7. Concomitant interventions/medications Locally. Dental or periodontal procedures, as required by the subject and as deemed necessary by the attending clinician, will be allowed before and during the trial.

Systemically. All necessary and not delayable concomitant interventions/medications will be allowed before and during the study. In case of incompatible concomitant systemic interventions/medications (e.g., bisphosphonates) assessed before the inclusion in the trial, the patient will not be included (see systemic exclusion criteria). In case the same treatments have been started after the patient inclusion but before the surgical treatment, the patient will be excluded from the trial (see "withdrawal criteria"). In case such treatments have been started after the surgical treatment, the patient will be retained in the study. Eventually, emergency medical care will always be allowed.

3.6. Statistical analysis

3.6.1. Sample Size Determination of the sample size was based on the mean deviation aft the implant platform between the static group and the dynamic group reported on previous studies: Putra et al., 2022, using the mean (SD) of the angular deviation between planned and implant insertion in G*Power (Version 3.1.9.7 software, Heinrich-Heine University, Dusseldorf, Germany). The effect size was estimated at 0.914, the significance level was set at 0,05 and the power at 0.80. The minimum required sample size resulted in 20 patients per group, but will be increased by 20%, expecting any possible dropouts. Thus, the final sample size will be adjusted to 48 patients, 24 in each group.

3.6.2. Statistical analysis Statistical analyses will be presented both at patient- and implant-level. Data will be reported as mean and SD unless otherwise specified (e.g., n [%]). Shapiro-Wilk goodness-of-fit test and histograms will be used to determine the normal distribution of the quantitative variables. Non-normally distributed variables will be additionally presented as medians and interquartile range (IQR). All analyses will be performed using the intention-to-treat population, and the last observation carried forward approach (LOCF) will be used for missing values.

The primary outcome will be accuracy as a compound parameter, where four different aspects will be measured: angular deviation, coronal deviation, apical deviation, and depth deviation. To assess the performance of the intervention, Students' t-test or Mann-Whitney U tests will be used for quantitative outcomes. Data on categorical outcomes will be compared using Chi-square test or Fisher-exact test. The secondary outcomes identified as relevant through the bivariant analysis will be included in a regression model, considering the accuracy as the primary outcome variable, which will be adjusted for confounding variables and factors such as the operators experience, type of surgical stent, etc.

Statistical significance will be set at p<0.05. The analysis will be performed using IBM SPSS Statistics (version 29.0.1.1, IBM Corporation, New York, NY, USA).

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients with one to four missing teeth, where dental implants are planned and where a tooth-supported or tooth-mucosal supported surgical guides can be fabricated. Free-ended situations will be allowed.
* Edentulous sites with at least 3 months of healing after tooth extraction.
* Staged hard and soft tissue augmentation will be permitted. In cases of previous bone augmentation (e.g. staged horizontal bone regeneration or lateral sinus lift), a minimum healing period of 6 months should be respected. In cases of previous soft tissue augmentation procedures, a minimum healing period of 2 months should be respected. Simultaneous close sinus lift procedures will be allowed when there is a minimum posterior bone height of 6 mm.
* Implants should be surrounded by at least 1.5 mm of bone.
* Periodontally healthy patients or with stable periodontal conditions after periodontal therapy. Periodontitis will be defined according to the EFP-AAP 2017 World Workshop Classification (Papapanou PN, Sanz M, et al., 2018): interdental CAL is detectable at ≥2 non-adjacent teeth or buccal or oral CAL ≥3 mm with pocketing ≥3 mm is detectable at ≥2 teeth, but the observed CAL cannot be ascribed to non-periodontitis-related causes such as 1) gingival recession of traumatic origin; 2) dental caries extending in the cervical area of the tooth; 3) the presence of CAL on the distal aspect of a second molar and associated with malposition or extraction of a third molar, 4) an endodontic lesion draining through the marginal periodontium; and 5) the occurrence of a vertical root fracture.
* Aged 21 years and over and able to sign an informed consent form.
* Enough available bone assessed on CBCT to place Klockner Vega implants of diameters ranging from 3.5 to 4.5 mm and lengths between 8 and 12 mm.

Exclusion Criteria:

1. Systemic

   * Completely edentulous patients or patients requiring mucosal- or bone-supported surgical guides.
   * Compromised general health (ASA IV-VI patients).
   * Systemic diseases which could influence the outcome of therapy (uncontrolled diabetes mellitus, bone disorders, etc.).
   * Pregnant or nursing women.
   * Chronic use of corticosteroids, nonsteroidal anti-inflammatory drugs (NSAID), or immune-modulator drugs (any type and dose).
   * Patients who need medications that affect bone metabolism (bisphosphonates, any type and dose).
   * Chronic diseases of the oral mucosa.
   * Smokers of >10 cigarettes/day.
   * >25% plaque index at the time of re-evaluation after non-surgical periodontal therapy and OHI
   * Unable to attend all study visits.
   * Need of simultaneous bone augmentation after implant placement to treat dehiscence and fenestration type defects or to augment bone contour (<1.5 mm of bone all around the implant circumference).
2. During surgery

   * Lack of primary stability assessed by hand testing after implant placement.
   * Less of 2 mm of keratinized mucosa, both at the lingual and buccal sites.
   * Lack of guide adjustment verified through the fitting windows.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-02-15 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Angular deviation | From planned implant position (presurgical digital plan) to final implant position (taken 3 months after implant placement, when performing the digital impression for the definitive crown)
  The discrepancy between the planned and actual placed implants will be measured to determine the accuracy of implant placement by superimposition of the virtual plan for the implant position and the postoperative scan. Angular deviation will be reported in degrees and will be measured from the most coronal point of the implant shoulder to the implant apex.
  All measurements will be performed by the same researcher, and in cases of more than one implant placed on the same patient the measurements will be performed separately. Measurements will be obtained digitally.

SECONDARY OUTCOMES:
Probing Depth (PD) | From the loading visit, to 6 and 12 month follow-up visits
  This measurement will be performed using a UNC15 calibrated plastic probe (Colorvue™, HuFriedy®, Chicago, IL, USA) at 6 sites per implant by a calibrated examiner at loading and 6- and 12-months visits.
  Defined as the distance in mm between the bottom of the probeable pocket and the margin of the peri-implant mucosa.
Bleeding on Probing (BoP) | From the loading visit, to 6 and 12 month follow-up visits
  This measurement will be performed using a UNC15 calibrated plastic probe (Colorvue™, HuFriedy®, Chicago, IL, USA) at 6 sites per implant by a calibrated examiner at loading and 6- and 12-months visits.
  Evaluated dichotomously as the presence or absence of bleeding within 15 seconds after gentle probing (about 20 g).
Suppuration on Probing (SUP) | From the loading visit, to 6 and 12 month follow-up visits
  This measurement will be performed using a UNC15 calibrated plastic probe (Colorvue™, HuFriedy®, Chicago, IL, USA) at 6 sites per implant by a calibrated examiner at loading and 6- and 12-months visits.
  Evaluated dichotomously as the presence or absence of suppuration after probing.
Keratinized Mucosa Width (KMW) | From the loading visit, to 6 and 12 month follow-up visits
  This measurement will be performed using a UNC15 calibrated plastic probe (Colorvue™, HuFriedy®, Chicago, IL, USA) at 6 sites per implant by a calibrated examiner at loading and 6- and 12-months visits.
  Measured as the distance in mm from the mid-buccal and mid-lingual mucosal margin to the mucosal junction.
Implant survival | 6 and 12 month follow up visits
  Implant survival will be evaluated at 6 months and 12 months after loading as the presence or absence of the implant over time.
Implant success | 6 and 12 month follow up visits
  Implant success will be defined as:
  * Absence of intraosseous implant mobility.
  * Absence of progressive marginal bone loss beyond expected physiologic remodeling.
  * Absence of structural implant failure.
Implant stability | During implant placement
  Implant stability will be assessed using Smart Pegs directly screwed to the implant connection at 10 Ncm to quantify implant stability quotient (ISQ) values.
Insertion torque | During implant placement
  During implant placement insertion torque will be measured by means of the motor handpiece.
Surgery difficulty | During implant placement
  The surgeon will answer on a 100-mm VAS scale just after the surgery to the following question: "How did you perceive the difficulty of the surgery?". The VAS scale will range from 0 (very simple) to 100 (very difficult).
Duration of surgery | During implant placement
  The time in minutes of the whole duration of the surgery, from the start of the anesthesia to the completion of the last suture.
Early Wound Healing | 2 weeks post-surgery
  The early wound healing will be evaluated at 2 weeks post-surgery. A modified Landry wound healing index will also be used, which assesses wound healing using scores ranging from 1 in a wound with a very poor healing index to a score of 5 representing excellent healing
Self Reported Pain | Immediately after surgery and 1-, 2-, 3-, 4-, 5-, 6-, 7 days post-operatively
  The patient will self-report on a 100-mm VAS scale ranging from 0 (no pain whatsoever) to 100 (worst pain imaginable) the perceived pain. The pain will be reported just after surgery and 1-, 2-, 3-, 4-, 5-, 6-, 7 days post-operatively in the evening, preferably at the same time.
Number of painkillers tablets | 1-, 2-, 3-, 4-, 5-, 6-, 7 days post-operatively
  The patient will document in the evening, preferably at the same time, the number and type of tablets taken each day from day-0 to day-7 post-surgery.
Swelling | Immediately after surgery and 1-, 2-, 3-, 4-, 5-, 6-, 7 days post-operatively
  The patient will self-report on a 100-mm VAS scale ranging from 0 (no swelling whatsoever) to 100 (worst swelling imaginable) the perceived swelling. The swelling will be reported just after surgery and 1-, 2-, 3-, 4-, 5-, 6-, 7 days post-operatively in the evening, preferably at the same time.
Discomfort during surgery | Immediately after surgery
  The patient will answer the following question on a 100-mm VAS scale just after the surgery: "How did you perceive the procedure?".
General patient satisfaction | 12-month visit
  The patient will self-report on a 100-mm VAS scale ranging from 0 to 100 overall satisfaction with the treatment received.
Radiographic marginal bone levels | Prosthetic loading visit (after loading of the prosthesis - which will be taken as the baseline measurement), 6 months after loading, and 12 months after loading.
  Standardized periapical digital radiographs will be taken the day of loading and at the 6- and 12-month visit after loading. Standardization will be assured using a custom-made bite block mounted on a film holder-beam aiming device (i.e., Rinn System [Dentsply International, York, PA, USA]) for each patient. A calibrated outcome assessor will perform the radiographic evaluation at the different time points to assess marginal bone levels (MBLs) at the mesial and distal aspect of each implant.
Interproximal emergence | Loading visit (14 weeks after implant placement - 12 weeks until impression, delivery 2 weeks after impression)
  The ideal emergence location of any implant is expected to be in the axis of the crown in a tooth-like form. An implant's emergence coinciding with interproximal tooth area is defined as a positioning error, it will be measure dichotomously after implant loading.
Insufficient inter-implant distance | Loading visit (14 weeks after implant placement - 12 weeks until impression, delivery 2 weeks after impression)
  For ease of hygiene and healthy maintenance of the surrounding tissues, a ≥2 mm distance is expected between any two neighbouring implants. A smaller distance is defined as a positioning error and will be measured dichotomously.
Excessive subcrestal placement | Loading visit (14 weeks after implant placement - 12 weeks until impression, delivery 2 weeks after impression)
  Implant shoulder platforms are expected to be 1-2 mm subcrestally. An implant's 3-mm or deeper shoulder level on the periapical x-ray is defined as a positioning error and will be measured dichotomously.
Implant-shoulder exposure | Loading visit (14 weeks after implant placement - 12 weeks until impression, delivery 2 weeks after impression)
  The whole body of the implant is expected to be not visible and surrounded by the bone and mucosa. An implant's body exposure in the shoulder area is defined as a positioning error, and will be measured dichotomously.
Improper screw access hole | Loading visit (14 weeks after implant placement - 12 weeks until impression, delivery 2 weeks after impression)
  Improper screw access hole. The access hole to the retention screw is expected to be on the occlusal surface. Any other position of the screw access hole is defined as a positioning error, and will be measured dichotomously.

CONTACTS AND LOCATIONS:
Overall Officials: Mariano Sanz, DDS, PHD, DrHC, Principal Investigator — Facultad de Odontología, Departamento de Especialidades Clínicas Odontológicas, Universidad Complutense de Madrid
Locations (1):
- Facultad de Odontología, Universidad Complutense de Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yi C, Li S, Wen A, Wang Y, Zhao Y, Zhang Y. Digital versus radiographic accuracy evaluation of guided implant surgery: an in vitro study. BMC Oral Health. 2022 Nov 24;22(1):540. doi: 10.1186/s12903-022-02585-5. PMID 36424579
- [Background] Younes F, Cosyn J, De Bruyckere T, Cleymaet R, Bouckaert E, Eghbali A. A randomized controlled study on the accuracy of free-handed, pilot-drill guided and fully guided implant surgery in partially edentulous patients. J Clin Periodontol. 2018 Jun;45(6):721-732. doi: 10.1111/jcpe.12897. Epub 2018 May 10. PMID 29608793
- [Background] Tang T, Liao L, Huang Z, Gu X, Zhang X. Accuracy of the evaluation of implant position using a completely digital registration method compared with a radiographic method. J Prosthet Dent. 2019 Dec;122(6):537-542. doi: 10.1016/j.prosdent.2018.11.020. Epub 2019 Apr 9. PMID 30979434
- [Background] Putra RH, Yoda N, Astuti ER, Sasaki K. The accuracy of implant placement with computer-guided surgery in partially edentulous patients and possible influencing factors: A systematic review and meta-analysis. J Prosthodont Res. 2022 Jan 11;66(1):29-39. doi: 10.2186/jpr.JPR_D_20_00184. Epub 2021 Jan 26. PMID 33504723
- [Background] Lo Russo L, Guida L, Mariani P, Ronsivalle V, Gallo C, Cicciu M, Laino L. Effect of Fabrication Technology on the Accuracy of Surgical Guides for Dental-Implant Surgery. Bioengineering (Basel). 2023 Jul 24;10(7):875. doi: 10.3390/bioengineering10070875. PMID 37508902
- [Background] Chai J, Liu X, Schweyen R, Setz J, Pan S, Liu J, Zhou Y. Accuracy of implant surgical guides fabricated using computer numerical control milling for edentulous jaws: a pilot clinical trial. BMC Oral Health. 2020 Oct 21;20(1):288. doi: 10.1186/s12903-020-01283-4. PMID 33087073
- [Background] Frizzera F, Calazans NNN, Pascoal CH, Martins ME, Mendonca G. Flapless Guided Implant Surgeries Compared with Conventional Surgeries Performed by Nonexperienced Individuals: Randomized and Controlled Split-Mouth Clinical Trial. Int J Oral Maxillofac Implants. 2021 Jul-Aug;36(4):755-761. doi: 10.11607/jomi.8722. PMID 34411217
- [Background] Abduo J, Lau D. Accuracy of static computer-assisted implant placement in anterior and posterior sites by clinicians new to implant dentistry: in vitro comparison of fully guided, pilot-guided, and freehand protocols. Int J Implant Dent. 2020 Mar 11;6(1):10. doi: 10.1186/s40729-020-0205-3. PMID 32157478
- [Background] Magrin GL, Rafael SNF, Passoni BB, Magini RS, Benfatti CAM, Gruber R, Peruzzo DC. Clinical and tomographic comparison of dental implants placed by guided virtual surgery versus conventional technique: A split-mouth randomized clinical trial. J Clin Periodontol. 2020 Jan;47(1):120-128. doi: 10.1111/jcpe.13211. Epub 2019 Nov 14. PMID 31628873
- [Background] Tattan M, Chambrone L, Gonzalez-Martin O, Avila-Ortiz G. Static computer-aided, partially guided, and free-handed implant placement: A systematic review and meta-analysis of randomized controlled trials. Clin Oral Implants Res. 2020 Oct;31(10):889-916. doi: 10.1111/clr.13635. Epub 2020 Jul 26. PMID 32654230
- [Background] Schwarz F, Ramanauskaite A. It is all about peri-implant tissue health. Periodontol 2000. 2022 Feb;88(1):9-12. doi: 10.1111/prd.12407. PMID 35103327
- [Background] Romandini M, Ruales-Carrera E, Sadilina S, Hammerle CHF, Sanz M. Minimal invasiveness at dental implant placement: A systematic review with meta-analyses on flapless fully guided surgery. Periodontol 2000. 2023 Feb;91(1):89-112. doi: 10.1111/prd.12440. Epub 2022 Jul 30. PMID 35906928
- [Background] Papaspyridakos P, Chen CJ, Singh M, Weber HP, Gallucci GO. Success criteria in implant dentistry: a systematic review. J Dent Res. 2012 Mar;91(3):242-8. doi: 10.1177/0022034511431252. Epub 2011 Dec 8. PMID 22157097
- [Background] Chackartchi T, Romanos GE, Parkanyi L, Schwarz F, Sculean A. Reducing errors in guided implant surgery to optimize treatment outcomes. Periodontol 2000. 2022 Feb;88(1):64-72. doi: 10.1111/prd.12411. PMID 35103317
- [Background] Albrektsson T, Wennerberg A. On osseointegration in relation to implant surfaces. Clin Implant Dent Relat Res. 2019 Mar;21 Suppl 1:4-7. doi: 10.1111/cid.12742. Epub 2019 Feb 28. PMID 30816639